CLINICAL TRIAL: NCT04979520
Title: A Small Pilot Study to Develop Biomarkers of Weekly Brodalumab Administration in Hidradenitis Suppurativa Patients
Brief Title: Molecular Characteristics of Brodalumab in Hidradenitis Suppurativa
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Principal Investigator, Yael Renert-Yuval, Instructor in clinical investigation, Rockefeller University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: YYU1014
Record Dates: First submitted 2021-07-09; First posted 2021-07-28 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Hidradenitis Suppurativa; Acne Inversa
Keywords: Hidradenitis Suppurativa; Acne Inversa; Brodalumab
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — brodalumab

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Brodalumab treated moderate-to-severe HS patients (Experimental): Weekly Brodalumab treatment 210mg/1.5ml, given subcutaneously for 12 weeks.
  Interventions: Drug: Brodalumab

INTERVENTIONS:
Drug: Brodalumab — Subcutaneously Brodalumab/Siliq, 210mg/1.5ml once a week
  Other Names: Siliq

SUMMARY:
Hidradenitis suppurativa is a disease involving skin folds, causing swelling of the skin and surrounding tissues, pain, and foul-smelling discharges. Effective treatment options are lacking. Recently, clinical trials conducted in our lab found Brodalumab was an effective drug for this disease. Weekly dosing achieved superior therapeutic outcomes compared to a dosing given once in every other week. Brodalumab was safe in both regimens, but blood and tissue studies to better understand this response are still needed. By performing this small pilot study and collecting blood and tissue samples from participants treated with Brodalumab once weekly we would like to better characterize the molecular response to this treatment, identify blood and tissue markers reflecting disease severity, and better understand disease mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical diagnosis of Hidradenitis Suppurativa by the Principal Investigator
* Age 18 to 99 years old
* Moderate to severe Hidradenitis Suppurativa with draining tunnels (Hidradenitis Suppurativa Severity Score System/IHS4>4)
* Must have medical insurance that is willing to pay for the study drug throughout the duration of the study

Exclusion Criteria:

* Inflammatory Bowel Disease
* HIV Positive
* Active Hepatitis B or C Infection
* Pregnant or Breastfeeding
* No concurrent use of any systemic antibiotics/retinoids/immunosuppressants/biologics (require washout period of >5 half-lives)
* A Score of >10 on the Beck's Depression Inventory (BDI) or on the Patient Health Questionnaire (PHQ)-9
* History of Keloid Scarring
* Any medical, psychological or social condition that, in the opinion of the Investigator, would jeopardize the health or well-being of the participant during any study procedures or the integrity of the data

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Interleukin-17 receptor A (IL-17RA) saturation during brodalumab administration at week 12 vs baseline | 12 weeks
  Percentage change in saturation

SECONDARY OUTCOMES:
Change in levels of IL-17A, IL-17C, IL-17, CXCL1, and CXCL8 | 12 weeks
  In Brodalumab treated participants at week 12 compared with baseline
Correlate IL-17R saturation (measured by the frequencies of immune cells positive to IL-17RA by flow cytometry) with clinical measures, such as pain or the Hidradenitis Suppurativa Severity Score System (IHS4) | 12 weeks
  In Brodalumab treated participants at week 12 compared with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Yael Renert-Yuval, MD, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No